CLINICAL TRIAL: NCT03324308
Title: The Safety, Feasibility and Accuracy of Dynamic Computed Tomography Myocardial Perfusion Imaging for Detection of Coronary Artery Disease
Brief Title: Dynamic Computed Tomography Myocardial Perfusion Imaging for Detection of Coronary Artery Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Redesign of Study.
Sponsor: Johns Hopkins University (Other)
Collaborators: Toshiba Medical Systems Corporation, Japan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00143208
Record Dates: First submitted 2017-10-17; First posted 2017-10-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Ischemia
Keywords: Coronary Artery Disease; Ischemia; Computed Tomography; Myocardial perfusion; Dynamic Imaging
MeSH Terms: conditions — Coronary Artery Disease; Ischemia | interventions — Computed Tomography Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional Group (Experimental): Participants undergoing dynamic computed tomography myocardial perfusion imaging.
  Intervention: Diagnostic Test: Dynamic Computed Tomography Angiography Imaging
  Interventions: Diagnostic Test: Computed Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Computed Tomography Angiography — This will be a prospective study comparing the low-dose dynamic vs. static CTP combined with the CTA for detecting hemodynamically significant coronary artery stenosis. Patients will have two 18-20 gauge intravenous lines placed for contrast administration. The following image sequences will be completed: coronary calcium scan (non-contrast), rest coronary arterial imaging (with 4-5 mL/sec intravenous ISOVUE-370 infusion), stress myocardial perfusion imaging 20 minutes after rest acquisition imaging (blood pressure will be checked then an infusion of adenosine will be started for a total of 5 minutes; after 5 minutes of adenosine infusion, CT perfusion imaging will be performed during a 4-5 mL/sec ISOVUE-370 infusion). Total estimated radiation dose: 10.551 mSv.
  Other Names: Myocardial Computed Tomography Perfusion - Static; Myocardial Computed Tomography Perfusion - Dynamic

SUMMARY:
Coronary artery computed tomographic angiography (CTA) is a widely used, highly accurate technique for the detection of coronary artery disease (CAD), with sensitivity and negative predictive values of over 90% (1-4). Patients with normal CTA findings have an excellent prognosis and do not require further testing for CAD (5). However, like invasive coronary angiography (QCA), CTA is an anatomic test and, unless lesions are very severe (>90% stenosis), cannot reliably predict the impairment of flow (functional significance) of intermediate grade stenoses.

For this reason, in approximately 15-25% of patients, additional functional testing may be required after CTA, usually in the form of stress testing (6-8). Stress testing is commonly done by exercise or pharmacologic stress with electrocardiographic monitoring and often, imaging of myocardial perfusion by nuclear scintigraphy (MPI) or detection of abnormal contraction by echocardiography. This requires a separate procedure, entailing time, expense and limited risk. Furthermore, in patients with previously known CAD, CTA alone is not an adequate test, because in most cases there are multiple lesions that are possible sources of ischemia.

Over the last 10 years, these investigators and others around the world have developed a method of imaging myocardial perfusion by CT (CTP). This test is an adjunct to the usual Cardiac Computed Tomography Angiography (CCTA) procedure and can be done immediately thereafter, using conventional pharmacologic stress agents. It has demonstrated accuracy in many single center trials, and in this large multicenter study, the CORE320 trial (9,10) which showed a high accuracy in predicting the combined results of QCA plus MPI testing and a second multicenter trial established non-inferiority of myocardial CTP compared with nuclear stress testing (11,12). Additionally, this investigator group has published a direct comparison of diagnostic performance of myocardial CTP imaging and SPECT myocardial perfusion imaging and demonstrated superior diagnostic performance of CTP imaging compared with SPECT for the diagnosis of significant disease on invasive angiography (13).

CTP images can be acquired with two different approaches: static or dynamic. In the CORE320 study, the CTP protocol used static acquisition method. The static CTP method, samples a snapshot of the iodine distribution in the blood pool and the myocardium over a short period of time, targeting either the upslope or the peak of contrast bolus. The notion behind this is that, at the upslope of the contrast, the difference in attenuation value of the ischemic and remote myocardium is at the maximum which enables for qualitative and semi-quantitative assessment of myocardial perfusion defects. The static CTP, however, does not allow for direct quantification of the myocardial blood flow (MBF). One of the drawbacks of static CTP lies in the acquirement of only one sample of data and the possibility of mistiming of the contrast bolus that results in poor contrast-to-tissue ratios by missing the peak attenuation (14). Output and flow rate of the contrast material may affect bolus timing. In addition, the acquisition of data from sequential heartbeats affects the attenuation gradient and may result in a heterogeneous iodine distribution, mimicking perfusion defects (15). Furthermore, the static CTP is limited in detection of balanced ischemia, where the perfusion of the entire myocardium is impaired and therefore there is no reference remote myocardium for comparison for semi-quantitative or qualitative static methods of CTP interpretation.

Dynamic CT perfusion imaging uses serial imaging over time to record the kinetics of iodinated contrast in the arterial blood pool and myocardium. This technique allows for multiple sampling of the myocardium and the blood pool and creating time attenuation curves (TAC) by measuring the change in CT attenuation over time. Mathematical modelling of TACs permits for direct quantification of MBF. Despite its advantages, the use of dynamic CTP were limited in the past. A high temporal resolution and high number of detectors are required for dynamic CTP to allow for entire myocardial coverage, and in order to obtain multiple consecutive images at high heart rates(16,17). But the main challenge of dynamic CTP acquisition was the high radiation dose associated with this technique. Nevertheless, with the introduction of the cutting-edge 320 detector CT scanning systems with fast gantry rotation the issue of the cardiac coverage is eliminated(17). The second-generation 320-row scanners also permit the quantification of the MBF with dynamic CTP acquisition with relatively low-dose of radiation(18,19).

In this study the investigators aim to evaluate the feasibility, safety and accuracy of the low-radiation dose dynamic myocardial CT perfusion compared to static CTP approach to detect hemodynamically significant coronary artery disease.

DETAILED DESCRIPTION:
This will be a prospective study comparing the low-dose dynamic vs. static CTP combined with the CTA for detecting hemodynamically significant coronary artery stenosis. The aim of the study is to assess the feasibility, safety and accuracy of low-dose dynamic CTP following CTA.

The study will enroll patients who have documented coronary artery disease and an indication for coronary angiography or CT angiography. Referred patients will be assessed for eligibility through phone calls followed by in-person interviews. Patents will be provided with the informed consent forms for CTA-CTP and iodine contrast if it is determined that participants are eligible for the study. Patients have the right to refuse to participate in the study and in that case participants will receive the regular care, per clinical guidelines. Baseline information will be collected from the patients after participants consent to participate in the study. Baseline data collection will happen at the same day that the patients will undergo CTA-CTP. The CTA-CTP acquisition takes less than 60 minutes after the patient is on the CT scanner table. Patient preparation time before patient is brought on the CT scanner depends on patients' heart rate and the time that takes to reduce patient's heart rate to a level that is appropriate for CTA-CTP acquisition. The blood sample will be obtained from the patients at the same day as CTA-CTP acquisition. Patients will be discharged to home at the same day participants undergo CTA-CTP.

b. Study duration and number of study visits required of research participants. There will be only one visit required for the purposes of the study, during which the CTA-CTP acquisition will be completed, baseline information will be collected and the blood samples will be drawn. The study participants will be contacted through phone 3-days after CTA-CTP acquisition for follow-up.

CT Imaging protocol

Patients will have two 18-20 gauge intravenous lines placed, one preferably in an antecubital vein for contrast administration. The patient will be hydrated with normal saline intravenously (250 - 500 ml) prior to CT scanning. The patient will lie supine on the scanner table and be attached to a 12 lead electrocardiographic monitor and an automated blood pressure monitor. Baseline ECG, heart rate, and blood pressure will be recorded and reviewed by one of the study investigators. Due to resultant artifacts from precordial leads, the 12 ECG leads and electrodes will be removed and rhythm monitoring will continue using the 3 lead system attached to the scanners monitoring system during scanning. A physician will be present at all times during adenosine infusion and CT imaging. Patients may receive an oral and/or intravenous dose of metoprolol up to one hour prior to the CT. If the heart rate is >60 beats per minute, 75 mg (max 80 mg) of metoprolol will be given orally. If Heart rate remains >60 beats per minute at the scan acquisition then, intravenous beta blocker (metoprolol, propranolol or landiolol) 2.5 - 5.0 mg every 5 minutes will be administered to achieve a heart rate between <60 beats per minute as blood pressure tolerates under the supervision of a physician. Scout images for determining scanning range will be obtained in the anterior-posterior and lateral views. Patients with systolic blood pressure ≥110 will receive sublingual fast acting short lasting nitrates (e.g. nitroglycerin, isosorbide dinitrate). Patients will then be asked to hold their breath (approximately 10-15 seconds) and non-contrast CT imaging will be performed starting just cranial to the coronary ostia and extending just caudal to the apex of the heart in order to obtain a coronary calcium score. CT angiogram will be performed to evaluate the coronaries and myocardial perfusion at rest. Blood pressure will be checked and intravenous adenosine infusion (0.14 mg/kg/min) will begin with continuous heart rate and rhythm monitoring. After 5 minutes of adenosine infusion, contrast-enhanced CT perfusion imaging will be performed during a 4-5 ml/sec intravenous iodinated contrast (ISOVUE®-370) infusion. Total contrast dose for the entire protocol will not exceed 140 ml and will be based on patient's body size. Patients will be asked to hold their breath during scanning. Immediately following completion of the scan, the adenosine infusion will be discontinued. A twelve lead ECG and blood pressure measurement will be repeated after discontinuation of adenosine and reviewed by a physician. Intravenous hydration will be continued during recovery with normal saline for a total volume for the entire post scan of 250 to 500 ml if deemed appropriate by the supervising physician.

320-Detector CT Protocol for Combined Coronary Angiography and Perfusion Imaging

1. Coronary calcium scan will be performed using the following protocol:

   * No contrast.
   * CT Imaging: tube voltage = 120kV, tube current = 140 Milliampere (mA), gantry rotation speed = 0.35 seconds, slice thickness = 0.5 mm, rows = 256-320, range = 128-160 mm. X-ray tube will be on for a total of 0.35 seconds. Estimated radiation dose = 1.5 Millisievert (mSv).
2. Rest coronary arterial imaging Rest perfusion and coronary arterial imaging will be performed during a 4-5 ml/sec intravenous iodinated contrast (ISOVUE®-370) infusion. The rest CTA-dynamic CTP images will be started using a test bolus acquisition and accurate quantification of optimum timing for dynamic CTP and boost CTA acquisition and will continue for 20-30 sec using a ECG triggering method to allow acquiring the images only within 70-80% of the R-R interval, but not continuously. The parameters for the dynamic CTP image acquisition are the followings: For the heart rate of <60 bpm the tube voltage will be 80 kV and the tube current will be 100mA. Other parameters are: gantry rotation=0.275, range=120mm. The CTA and static CTP imaging will be performed as a boost scan during the dynamic CTP with the same tube voltage (80kV) but the tube current of 600mA within 70-80% of R-R interval. The boost timing will be quantified from test bolus acquisition. The average radiation dose for rest CTA and rest dynamic and static CTP acquisition is 3.69mSv.
3. Stress Myocardial Perfusion imaging 20 minutes after rest image acquisition Blood pressure will be checked and intravenous adenosine infusion will begin with continuous heart rate and rhythm monitoring. After 5 minutes of adenosine infusion, contrast-enhanced CT perfusion imaging will be performed during a 4-5 ml/sec intravenous iodinated contrast (ISOVUE®-370) infusion. The stress dynamic CTP images will be started using a test bolus acquisition and accurate quantification of optimum timing for dynamic CTP and boost CTA acquisition and will continue for 20-30 sec using a ECG triggering method to allow acquiring the images only within 70-80% of the R-R interval, but not continuously. The parameters for the stress dynamic CTP image acquisition are the followings: For the heart rate of <80 bpm the tube voltage will be 80 kV and the tube current will be 100mA. Other parameters are: gantry rotation=0.275, range=120mm. The stress static CTP imaging will be performed as a boost scan during the stress dynamic CTP with the same tube voltage (80kV) but the tube current of 600mA within 70-80% of R-R interval. The boost timing will be quantified from test bolus acquisition. The average radiation dose for stress dynamic and static CTP acquisition is 5.17mSv.

The estimated average radiation dose for the entire cardiac computed protocol is 10.55 mSv and shall not exceed 15mSv. Beta-blockers will be used to control the heart rate and thus maintain the radiation dose as low as reasonably achievable. The total contrast dose will not exceed 140 ml. Depending on patient size, 50-70 ml of iodinated contrast will be used for each of rest and stress scans.

In the event that the CT raw data are not readable at the Johns Hopkins University, a copy of the raw data (anonymized without patient identifiers) will be transferred to Toshiba Medical Systems for engineering support of image reconstruction in these isolated cases. Toshiba Medical Systems will perform the image reconstruction and return the raw data and the reconstructed image data to the Johns Hopkins University for image analysis.

Within 3 weeks of the CT, the CT will be reviewed for non-cardiac findings by a locally qualified, institutionally approved cardiologist and reported to the patient's clinical physician and patient in a timely fashion preferably prior to or during the 30-day follow-up.

c. Blinding, including justification for blinding or not blinding the trial, if applicable.

Dynamic and static CTP images will be analyzed separately and when analyzing the CTP images with each method, the readers will be blinded to the results the other method. However the readers will have access to the results for CTA interpretation while reading the CTP images with either of static or dynamic methods.

d. Justification of why participants will not receive routine care or will have current therapy stopped.

The study will be only enrolling patients with an indication for CTA or invasive coronary angiography and will undergo these tests. So routine care will be delivered to the participants.

7. Study Statistics

a. Primary outcome variable. The primary outcome measures will be feasibility, safety and accuracy of dynamic CTP-CTA compared to static CTP-CTA to detect hemodynamically significant coronary artery stenosis. The hemodynamically significant coronary artery stenosis will be defined as having at least one vessel with a ≥50% stenosis associated with perfusion defect in static CTP images.

At the index visit, failure to complete the CTP protocol will constitute an incomplete study and such patients will be excluded from the per protocol analysis. All patients completing the CTP protocol and providing informed consent will be included in per-protocol analyses. All data from all consented patients who do not complete the CTP protocol will be included in the intent-to-diagnose analysis.

Descriptive statistics will be given for all variables including indications for the test, demographics, patient history, CTA test information, dynamic and static CTP information. Categorical variables will be summarized as counts and percentages. All continuous variables will be summarized as means+/- the standard deviation followed by the median, minimum and maximum and 25th, 75th percentiles where needed.

The frequency of the primary safety outcomes [death, myocardial infarction, unstable angina, ventricular tachycardia, asystole, severe bradycardia, allergic skin reactions, allergic respiratory reactions, hypotension, anaphylaxis and contrast induced nephropathy] will all be summarized; 95% binomial confidence intervals for the proportions of these outcomes will be calculated. The additional safety outcomes involving CTP complications will be summarized with frequencies and 95% confidence intervals for proportions. Radiation dose and efficiency measures (duration(s) involving the CTP procedure) will be summarized overall with median and 25th and 75th percentiles. Also minima and maxima will be provided. The investigators may explore possible associations between patient characteristics [demographics (gender, age), prior histories or indications] and the binary safety outcomes using contingency table methods, t tests or Wilcoxon Rank Sum, as appropriate. Associations between radiation dose and patient characteristics may be explored with nonparametric methods. The investigators may also explore possible relationships between the CTA stenosis categories (0%, 1-49%, 50-100%) and the dynamic and static CTP results. The occurrence of clinical events recorded at 30-day chart review will be related to the category of CTP final results (Normal, Probably Normal, Equivocal, Probably Abnormal and Abnormal) using methods for contingency tables which incorporate the natural ordering of CTP categories.

The frequency of the studies with the adequate image quality for interpretation of dynamic CTP images will be reported as a measure is feasibility. This feasibility index will be also reported at the myocardial segment level and the frequency of Left Ventricular (LV) segments with adequate dynamic CTP image quality will be reported.

The inter- and intra-reader reproducibility of dynamic CTP interpretation will be assessed using kappa statistics, intra-class correlation coefficients and Bland-Altman plot, as appropriate.

The accuracy of the dynamic CTP for detection of hemodynamically significant coronary artery stenosis will be based on the area under the receiver operating characteristic (ROC) curve (AUC) with the static CTP results as the comparator. The correlation of the dynamic vs. static CTP will be also assessed in the categorical (Chi-squared test) and continuous (Spearman's correlation coefficient) scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for invasive coronary angiography or CT angiography
* Documented coronary artery disease defined as presence of one or more of the following:
* CAD documented by invasive coronary angiography or CT angiography
* History of typical stable angina and receiving guideline-driven therapy for coronary artery disease for ≥ 1 month prior to consent
* History of hospitalization for unstable angina with no active acute coronary syndrome within 48 hours prior to scan
* Refractory angina defined as marked limitation of ordinary physical activity or inability to perform ordinary physical activity without discomfort, with an objective evidence of myocardial ischemia and persistence of symptoms despite optimal medical therapy, life style modification treatments, and revascularization therapies
* Able to understand and willing to sign the Informed Consent Form.

Exclusion Criteria:

* Known allergy to iodinated contrast media
* History of contrast-induced nephropathy
* History of multiple myeloma or previous organ transplantation
* Elevated serum creatinine (> 1.5mg/dl) OR calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula)
* Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block)
* Evidence of severe symptomatic heart failure (NYHA Class III or IV); Known or suspected moderate or severe aortic stenosis
* Previous coronary artery bypass or other cardiac surgery
* Coronary artery intervention (PCI) within the last 6 months
* Known or suspected intolerance or contraindication to beta-blockers including:
* Known allergy to beta-blockers
* History of moderate to severe bronchospastic lung disease (including moderate to severe asthma)
* Severe pulmonary disease (chronic obstructive pulmonary disease) with the use of inhaled bronchodilators over the past year
* Presence of any other history or condition that the investigator feels would be problematic
* History of high radiation exposure defined as ≥2 nuclear or CT studies or ≥ 5.0 reml within 18 months prior to the scan
* Does the patient have active acute coronary syndrome within 48 hours prior to consent?

  * Typical, prolonged (>20 minute) rest angina at admission
  * Angina equivalent symptoms compatible with ischemia plus abnormal cardiac enzymes
  * Prolonged rest chest pain (>20 minutes) resolved before admission plus prior ischemic ECG changes
  * Rest chest pain < 20 minutes relieved with nitrates in the prior 48 hours plus prior ischemic ECG changes.
  * If yes to any of the above, Calculate Thrombolysis in Myocardial Infarction (TIMI) risk score:

    * If TIMI risk score ≥ 5 OR elevated cardiac enzymes in the 72 hours prior patient is excluded.
    * If TIMI risk score is <5 and cardiac enzymes are normal patient is included.
  * If all of above are no then patient is included.
* Implantable cardioverter-defibrillator (but not pacemakers) within the imaging field of view
* Contraindications to vasodilator stress agents:

  * Systolic Blood Pressure (SBP)<90mmHg, -Recent use of dipyridamole and dipyridamole containing medications - -Recent use of methylxanthines (aminophylline and caffeine) - -Unstable acute Myocardial Infarction (MI) or acute coronary syndrome -
  * Profound sinus bradycardia (<40 bpm)
* Body Mass Index greater than 30

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety and tolerability) | 30 days post procedure
  Occurrence of treatment emergent adverse events including allergic reactions, adverse reactions to pharmacologic stress agents, contrast induced nephropathy

SECONDARY OUTCOMES:
The Area Under Receiver Operating Characteristics Curve (AUC) of combined CTA-dynamic CTP for detection of hemodynamically significant coronary artery stenosis at the patient level | At the day of procedure
  At the patient level: The Area Under Receiver Operating Characteristics Curve (AUC) of combined CTA-dynamic CTP for detection of hemodynamically significant coronary artery stenosis by combined CTA-static CTP defined as at least one vessel with ≥50% stenosis with an associated perfusion defect in static CTP.
The Area Under Receiver Operating Characteristics Curve (AUC) of dynamic CTP for detection of a perfusion defect at the patient level | At the day of procedure
  At the patient level: The Area Under Receiver Operating Characteristics Curve (AUC) of dynamic CTP for detection of a perfusion defect compared to static CTP.
The Area Under Receiver Operating Characteristics Curve (AUC) of combined CTA-dynamic CTP for detection of hemodynamically significant coronary artery stenosis at the vessel level. | At the day of procedure
  At the vessel level: The Area Under Receiver Operating Characteristics Curve (AUC) of combined CTA-dynamic CTP for detection of hemodynamically significant coronary artery stenosis by combined CTA-static CTP defined a coronary artery lesion with ≥50% stenosis with an associated perfusion defect in the same artery in static CTP.
The Area Under Receiver Operating Characteristics Curve (AUC) of dynamic CTP for detection of a perfusion defect at the vessel level. | At the day of procedure
  At the vessel level: The Area Under Receiver Operating Characteristics Curve (AUC) of dynamic CTP for detection of a perfusion defect compared to static CTP.
Total length of stay (hours) | 1-7 days after the procedure
  Total length of stay including hospital stay if admitted (hours).
Duration of exam (hours) | 24 hours after initiation of exam
  Time from initiation to completion of CCTA and CTP testing (hours)
Interpretation time (hours) | 1-4 hours after initiation of test interpretation
  Time to interpret the test (hours)
Frequency of interpretable images | At the day of procedure
  Frequency of the studies with the adequate image quality for interpretation of dynamic CTP images
Frequency of interpretable myocardial segments | At the day of procedure
  Frequency of the myocardial segments with adequate dynamic CTP image quality for interpretation
The inter-reader reproducibility of dynamic CTP image interpretation | 1-7 days after the exam
  The inter-reader reproducibility of dynamic CTP image interpretation using Concordance Correlation Coefficient
The intra-reader reproducibility of dynamic CTP image interpretation | 1-7 days after the exam
  The intra-reader reproducibility of dynamic CTP image interpretation using Concordance Correlation Coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Unversity School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Hamon M, Biondi-Zoccai GG, Malagutti P, Agostoni P, Morello R, Valgimigli M, Hamon M. Diagnostic performance of multislice spiral computed tomography of coronary arteries as compared with conventional invasive coronary angiography: a meta-analysis. J Am Coll Cardiol. 2006 Nov 7;48(9):1896-910. doi: 10.1016/j.jacc.2006.08.028. Epub 2006 Sep 26. PMID 17084268
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] Abdulla J, Asferg C, Kofoed KF. Prognostic value of absence or presence of coronary artery disease determined by 64-slice computed tomography coronary angiography a systematic review and meta-analysis. Int J Cardiovasc Imaging. 2011 Mar;27(3):413-20. doi: 10.1007/s10554-010-9652-x. Epub 2010 Jun 12. PMID 20549366
- [Background] Gallagher MJ, Ross MA, Raff GL, Goldstein JA, O'Neill WW, O'Neil B. The diagnostic accuracy of 64-slice computed tomography coronary angiography compared with stress nuclear imaging in emergency department low-risk chest pain patients. Ann Emerg Med. 2007 Feb;49(2):125-36. doi: 10.1016/j.annemergmed.2006.06.043. Epub 2006 Sep 15. PMID 16978738
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Goldstein JA, Chinnaiyan KM, Abidov A, Achenbach S, Berman DS, Hayes SW, Hoffmann U, Lesser JR, Mikati IA, O'Neil BJ, Shaw LJ, Shen MY, Valeti US, Raff GL; CT-STAT Investigators. The CT-STAT (Coronary Computed Tomographic Angiography for Systematic Triage of Acute Chest Pain Patients to Treatment) trial. J Am Coll Cardiol. 2011 Sep 27;58(14):1414-22. doi: 10.1016/j.jacc.2011.03.068. PMID 21939822
- [Background] George RT, Arbab-Zadeh A, Cerci RJ, Vavere AL, Kitagawa K, Dewey M, Rochitte CE, Arai AE, Paul N, Rybicki FJ, Lardo AC, Clouse ME, Lima JA. Diagnostic performance of combined noninvasive coronary angiography and myocardial perfusion imaging using 320-MDCT: the CT angiography and perfusion methods of the CORE320 multicenter multinational diagnostic study. AJR Am J Roentgenol. 2011 Oct;197(4):829-37. doi: 10.2214/AJR.10.5689. PMID 21940569
- [Background] Rochitte CE, George RT, Chen MY, Arbab-Zadeh A, Dewey M, Miller JM, Niinuma H, Yoshioka K, Kitagawa K, Nakamori S, Laham R, Vavere AL, Cerci RJ, Mehra VC, Nomura C, Kofoed KF, Jinzaki M, Kuribayashi S, de Roos A, Laule M, Tan SY, Hoe J, Paul N, Rybicki FJ, Brinker JA, Arai AE, Cox C, Clouse ME, Di Carli MF, Lima JA. Computed tomography angiography and perfusion to assess coronary artery stenosis causing perfusion defects by single photon emission computed tomography: the CORE320 study. Eur Heart J. 2014 May;35(17):1120-30. doi: 10.1093/eurheartj/eht488. Epub 2013 Nov 19. PMID 24255127
- [Background] Cury RC, Kitt TM, Feaheny K, Blankstein R, Ghoshhajra BB, Budoff MJ, Leipsic J, Min JK, Akin J, George RT. A randomized, multicenter, multivendor study of myocardial perfusion imaging with regadenoson CT perfusion vs single photon emission CT. J Cardiovasc Comput Tomogr. 2015 Mar-Apr;9(2):103-12.e1-2. doi: 10.1016/j.jcct.2015.01.002. Epub 2015 Jan 7. PMID 25726411
- [Background] Cury RC, Kitt TM, Feaheny K, Akin J, George RT. Regadenoson-stress myocardial CT perfusion and single-photon emission CT: rationale, design, and acquisition methods of a prospective, multicenter, multivendor comparison. J Cardiovasc Comput Tomogr. 2014 Jan-Feb;8(1):2-12. doi: 10.1016/j.jcct.2013.09.004. Epub 2013 Oct 18. PMID 24314823
- [Background] George RT, Mehra VC, Chen MY, Kitagawa K, Arbab-Zadeh A, Miller JM, Matheson MB, Vavere AL, Kofoed KF, Rochitte CE, Dewey M, Yaw TS, Niinuma H, Brenner W, Cox C, Clouse ME, Lima JA, Di Carli M. Myocardial CT perfusion imaging and SPECT for the diagnosis of coronary artery disease: a head-to-head comparison from the CORE320 multicenter diagnostic performance study. Radiology. 2014 Aug;272(2):407-16. doi: 10.1148/radiol.14140806. Epub 2014 May 26. PMID 24865312
- [Background] Bischoff B, Bamberg F, Marcus R, Schwarz F, Becker HC, Becker A, Reiser M, Nikolaou K. Optimal timing for first-pass stress CT myocardial perfusion imaging. Int J Cardiovasc Imaging. 2013 Feb;29(2):435-42. doi: 10.1007/s10554-012-0080-y. Epub 2012 Jun 20. PMID 22714549
- [Background] Danad I, Szymonifka J, Schulman-Marcus J, Min JK. Static and dynamic assessment of myocardial perfusion by computed tomography. Eur Heart J Cardiovasc Imaging. 2016 Aug;17(8):836-44. doi: 10.1093/ehjci/jew044. Epub 2016 Mar 24. PMID 27013250
- [Background] Schuleri KH, George RT, Lardo AC. Applications of cardiac multidetector CT beyond coronary angiography. Nat Rev Cardiol. 2009 Nov;6(11):699-710. doi: 10.1038/nrcardio.2009.172. PMID 19851349
- [Background] Valdiviezo C, Ambrose M, Mehra V, Lardo AC, Lima JA, George RT. Quantitative and qualitative analysis and interpretation of CT perfusion imaging. J Nucl Cardiol. 2010 Dec;17(6):1091-100. doi: 10.1007/s12350-010-9291-6. PMID 20924735
- [Background] Kikuchi Y, Oyama-Manabe N, Naya M, Manabe O, Tomiyama Y, Sasaki T, Katoh C, Kudo K, Tamaki N, Shirato H. Quantification of myocardial blood flow using dynamic 320-row multi-detector CT as compared with (1)(5)O-H(2)O PET. Eur Radiol. 2014 Jul;24(7):1547-56. doi: 10.1007/s00330-014-3164-3. Epub 2014 Apr 18. PMID 24744200
- [Background] Fujita M, Kitagawa K, Ito T, Shiraishi Y, Kurobe Y, Nagata M, Ishida M, Sakuma H. Dose reduction in dynamic CT stress myocardial perfusion imaging: comparison of 80-kV/370-mAs and 100-kV/300-mAs protocols. Eur Radiol. 2014 Mar;24(3):748-55. doi: 10.1007/s00330-013-3063-z. Epub 2013 Nov 22. PMID 24272224
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):485-510. doi: 10.1016/j.jacc.2012.11.018. Epub 2012 Dec 17. No abstract available. PMID 23256913
- [Background] Jneid H, Anderson JL, Wright RS, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP. 2012 ACCF/AHA focused update of the guideline for the management of patients with unstable angina/non-ST-elevation myocardial infarction (updating the 2007 guideline and replacing the 2011 focused update): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2012 Aug 14;60(7):645-81. doi: 10.1016/j.jacc.2012.06.004. Epub 2012 Jul 16. No abstract available. PMID 22809746
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO, Tracy CM, Epstein AE, Darbar D, DiMarco JP, Dunbar SB, Estes NA 3rd, Ferguson TB Jr, Hammill SC, Karasik PE, Link MS, Marine JE, Schoenfeld MH, Shanker AJ, Silka MJ, Stevenson LW, Stevenson WG, Varosy PD; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Heart Rhythm Society. 2012 ACCF/AHA/HRS focused update incorporated into the ACCF/AHA/HRS 2008 guidelines for device-based therapy of cardiac rhythm abnormalities: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2013 Jan 22;61(3):e6-75. doi: 10.1016/j.jacc.2012.11.007. Epub 2012 Dec 19. No abstract available. PMID 23265327
- [Background] George RT, Silva C, Cordeiro MA, DiPaula A, Thompson DR, McCarthy WF, Ichihara T, Lima JA, Lardo AC. Multidetector computed tomography myocardial perfusion imaging during adenosine stress. J Am Coll Cardiol. 2006 Jul 4;48(1):153-60. doi: 10.1016/j.jacc.2006.04.014. Epub 2006 Jun 21. PMID 16814661
- [Background] Schwarz F, Hinkel R, Baloch E, Marcus RP, Hildebrandt K, Sandner TA, Kupatt C, Hoffmann V, Wintersperger BJ, Reiser MF, Theisen D, Nikolaou K, Bamberg F. Myocardial CT perfusion imaging in a large animal model: comparison of dynamic versus single-phase acquisitions. JACC Cardiovasc Imaging. 2013 Dec;6(12):1229-38. doi: 10.1016/j.jcmg.2013.05.018. Epub 2013 Oct 23. PMID 24269264
- [Background] Bamberg F, Becker A, Schwarz F, Marcus RP, Greif M, von Ziegler F, Blankstein R, Hoffmann U, Sommer WH, Hoffmann VS, Johnson TR, Becker HC, Wintersperger BJ, Reiser MF, Nikolaou K. Detection of hemodynamically significant coronary artery stenosis: incremental diagnostic value of dynamic CT-based myocardial perfusion imaging. Radiology. 2011 Sep;260(3):689-98. doi: 10.1148/radiol.11110638. PMID 21846761
- [Background] Ishida M, Kitagawa K, Ichihara T, Natsume T, Nakayama R, Nagasawa N, Kubooka M, Ito T, Uno M, Goto Y, Nagata M, Sakuma H. Underestimation of myocardial blood flow by dynamic perfusion CT: Explanations by two-compartment model analysis and limited temporal sampling of dynamic CT. J Cardiovasc Comput Tomogr. 2016 May-Jun;10(3):207-14. doi: 10.1016/j.jcct.2016.01.008. Epub 2016 Jan 13. PMID 26851149
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441